CLINICAL TRIAL: NCT00572312
Title: Influence of Adding Atorvastatin to Dual Renin-Angiotensin-Aldosterone System Blockade on Proteinuria
Brief Title: Optimalization of Nephroprotection Using Atorvastatin (Sortis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ST-4/ATOR/01
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Chronic Kidney Disease; Proteinuria
Keywords: Proteinuria,; atorvastatin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin (Sortis) 40 mg — In the 8-weeks run-in period angiotensin-converting enzyme inhibitors and angiotensin II type 1 receptor blockers were administered to achieve the target blood pressure below 130/80 mmHg. Next, they were randomly assigned to add (or not) 40 mg of atorvastatin in two active treatment periods lasting 8 weeks each

SUMMARY:
The main purpose of the study is find whether the addition of statin (Atorvastatin) to dual renin-angiotensin-aldosterone system blockade involving angiotensin converting enzyme inhibitor and AT-1 angiotensin II receptor blocker leads to the reduction of proteinuria, main prognostic marker of chronic kidney disease progression.

DETAILED DESCRIPTION:
The renin-angiotensin-aldosterone system (RAAS) plays an important role in the progression of chronic kidney diseases (CKD), and inhibition of the RAAS with angiotensin-converting enzyme inhibitors (ACEI) and angiotensin II type 1 receptor blockers (ARB) may retard CKD progression. Dual pharmacological blockade of the RAAS with ACEI and ARB is recommended as a standard renoprotective management at least in patients with nondiabetic proteinuric CKD. However, neither ACEI nor ARB, even in high doses or in concomitant usage, abrogate the progression of CKD completely. Innovative approaches are needed to keep patients with CKD off dialysis. Additional statin (Atorvastatin) pathway may prove to be such beneficial therapeutic concept.Given these facts additional administration of statin to combination treatment with ACEI and ARB, may provide additional renal protection. To shed more light on this issue, we performed a randomised open controlled study to evaluate the influence of triple therapy with ACEI and/orARB and statin on surrogate markers of kidney injury, i.e. proteinuria, markers of tubular involvement and kidney fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Stable proteinuria above 300 mg/24 hours (no variations above 25% in the last 6 months)
* Normal or slightly impaired stable renal function defined as serum creatinine level below 1.7 mg/dl (eGFR > 45 ml/min)

Exclusion Criteria:

* Nephrotic syndrome
* Steroids or other immunosuppressive treatment minimum during six months before the study
* Diabetes mellitus
* Potassium serum level > 5.1 mEq/L
* Albumin serum level < 2.0mg/dL
* Creatinine serum level >2 mg/dl
* Current diagnosis of heart failure New York Heart Association (NYHA) Class II-IV
* Clinically significant valvular heart disease or second or third degree heart block without a pacemaker
* History of hypertensive encephalopathy, cerebrovascular accident or transient ischemic cerebral attack
* History of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any percutaneous coronary intervention
* History of malignancy including leukemia and lymphoma (but not basal cell skin carcinoma) within the past five years
* Pregnant or nursing women
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs.
* History of alcohol abuse
* NSAID abuse (more than 2 doses per week)
* Known or suspected contraindications to the study medications, including history of allergy to ACE inhibitors, AT-1 receptor blockers and atorvastatin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02

PRIMARY OUTCOMES:
Investigate the antiproteinuric effect of adding atorvastatin to the combination therapy with angiotensin converting enzyme inhibitor and AT-1 receptor blocker in maximal recommended doses

SECONDARY OUTCOMES:
Investigate the effect of the study intervention on urine excretion of N-acetyl-β-D-glucosaminidase, alfa1-microglobulin and amino-terminal propeptide of type III procollagen.

CONTACTS AND LOCATIONS:
Overall Officials: Boleslaw Rutkowski, MD PhD, Principal Investigator — Department of Nephrology Transplantology and Internal Medicine. Medical University of Gdansk.

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702